CLINICAL TRIAL: NCT00714610
Title: Serum Metal Ion Concentrations Following Unilateral Versus Bilateral Large Head Metal on Metal Primary Hip Arthroplasty
Brief Title: Serum Metal Ion Concentrations Following Primary Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Peters, M.D., University of Utah
Other Study IDs: 21498
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Serum metal ion concentration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood will be drawn for analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Unilateral or bilateral large head metal on metal primary total hip arthroplasty

SUMMARY:
The objective of this study is to compare serum chromium and cobalt levels of patients who have undergone metal on metal total hip arthroplasty. It is unknown if the presence of bilateral well-functioning large-head metal-on-metal (MOM) total hip arthroplasties (THAs) leads to higher serum metal ion concentrations than unilateral MOM THA. Elevated levels (chromium, 17 μg/L; cobalt, 19 μg/L) have been associated with poorly functioning MOM THA with metallosis. Fourteen patients having undergone bilateral and 25 patients having undergone unilateral large-head primary MOM THA were compared. Harris Hip Scores, University of California Los Angeles activity scores, radiographs, serum creatinine, and serum cobalt and chromium levels were obtained.

DETAILED DESCRIPTION:
The objective of this study is to compare serum chromium and cobalt levels of patients who have undergone metal on metal total hip arthroplasty.

The effect of the presence of bilateral large-head MOM THA on circulating metal ions levels has not been thoroughly studied. Metal ion levels in patients with unilateral MOM vs bilateral MOM resurfacing and small-head THA have been reported; however, to the investigators knowledge, no study has investigated the differences in serum metal ion levels in unilateral vs bilateral largehead (≥38 mm) MOM THA. The objective of this study was to compare serum cobalt and chromium levels in patients who have undergone unilateral vs bilateral large-head MOM THA to better understand the effect of the presence of bilateral implants on circulating metal ion levels. The investigators believe that further understanding baseline levels in well-functioning MOM THA will increase the clinical utility of checking serum metal ion levels in the workup of the painful MOM THA. The investigators hypothesis was that serum metal ion levels in patients with well-functioning bilateral large-head MOM THA would be higher than levels in patients with well functioning unilateral large-head MOM THA, but these levels would not approach those seen with metallosis.

ELIGIBILITY:
Inclusion Criteria:

* undergone unilateral large-head (≥38 mm) primary MOM THA
* undergone bilateral large-head primary MOM THA
* 18 years old or older
* at least one year out from their index procedure
* had well-positioned components

Exclusion Criteria:

* other metal implants
* renal insufficiency (estimated creatinine clearance b30 mL/min)
* component malpositioning (cup inclination angle N55°)
* evidence of osteolysis on radiographs
* a poorly functioning hip (Harris Hip Score [HHS] b70)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups were identified: the first group having undergone unilateral large-head (≥38 mm) primary MOM THA and the second having undergone bilateral large-head primary MOM THA. Patients were at least 18 years old, were at least 1 year out from their index procedure, and had well-positioned components.
  Patients in both cohorts had cementless modular titanium alloy proximally porous-coated, tapered femoral stems (Biomet Taperloc or Bi-Metric; Biomet, Warsaw, Ind).
  All surgeries were done between the years of 2003 and 2009.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Serum Metal Ion Concentrations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Peters, MD, Principal Investigator — University of Utah Orthopaedic Center
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States